CLINICAL TRIAL: NCT05037435
Title: Prospective, Randomized, Double-blind, Placebo-controlled Clinical Study of the Safety and Efficacy of the Vaccine for the Prevention of Pentavalent Live Rotavirus Infection in Healthy Subjects (Target Age of 18-45 Years Old).
Brief Title: Safety and Immunological Efficacy of the Pentavalent Rotavirus Vaccine - Rota-V-Aid™ (Live Attenuated Oral, Freeze-dried) at Healthy Adults Aged 18 to 45 Years.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Limited Liability Company Pharm Aid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: RTB 001/18
Record Dates: First submitted 2021-08-18; First posted 2021-09-08 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Rotavirus Infections; Rotavirus Vaccines
MeSH Terms: conditions — Rotavirus Infections | interventions — Freeze Drying

STUDY DESIGN:
Intervention Model Description: Prospective randomized double-blind placebo-controllable.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The pentavalent rotavirus vaccine - Rota-V-Aid™ (live attenuated oral, freeze-dried) (Experimental): Live attenuated bovine-human [UK] reassortant rotavirus vaccine manufactured by the Serum Institute of India, Limited (SIIL). The pentavalent vaccine contains rotavirus serotypes G1, G2, G3, G4, and G9 (≥5.6 log10 FFU/serotype/dose). The vaccine is lyophilized and supplied with 2.5 ml of citrate bicarbonate buffer added for reconstitution before oral administration.
  Interventions: Biological: The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried)
- Diluent is a sterile solution (Citrate Bicarbonate Buffer) (Placebo Comparator): Same constituents as the active vaccine but without the viral antigens; manufactured by SIIL.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: The pentavalent rotavirus vaccine (live attenuated oral, freeze-dried) — Group 1 (20 participants) - received the pentavalent live vaccine to prevent rotavirus infection Single-use orally 2.5 ml (1 dose).
  Other Names: Rota-V-Aid™
  Arms: The pentavalent rotavirus vaccine - Rota-V-Aid™ (live attenuated oral, freeze-dried)
Other: Placebo — Group 2 (20 participants ) - received placebo orally once of 2.5 ml (1 dose).
  Other Names: Diluent is a sterile solution (Citrate Bicarbonate Buffer)
  Arms: Diluent is a sterile solution (Citrate Bicarbonate Buffer)

SUMMARY:
The purpose of the presented study was to evaluate the safety and immunological efficacy in preventing the rotavirus infection within a cohort of healthy subjects (target age of 18-45 years old) by using the pentavalent rotavirus vaccine - Rota-V-Aid™ (live attenuated oral, freeze-dried).

DETAILED DESCRIPTION:
The clinical study named "Prospective, randomized, double-blind, placebo-controlled study of safety and immunological efficacy for preventing a rotavirus infection pentavalent vaccine, live attenuated at the healthy subjects at the age of 18-45 years" was conducted in the Russian Federation. The mentioned study was performed as per Protocol of clinical trial No. RTB 001/18 (given by MOH RF exp June 7, 2018). All relevant requirements of the National Legislative system and the international rules of conduct of clinical trials (ICH GCP).

The study objective was to assess the safety and immunological efficacy for preventing a rotavirus infection pentavalent rotavirus vaccine - Rota-V-Aid™ (live attenuated oral, freeze-dried) at healthy adults aged 18 to 45 years for the subsequent vaccination of the children's contingent.

For the achievement of a goal, it was necessary to solve the following problems:

1. Assessment of the vaccine's safety for preventing a rotavirus infection pentavalent live compared to placebo at a single oral introduction to volunteers at the age of 18-45 years.
2. Immunological efficacy assessment for prevention of a rotavirus infection pentavalent live in comparison with placebo at a single oral introduction to volunteers at the age of 18-45 years

ELIGIBILITY:
Inclusion Criteria:

1. The signed informed consent;
2. Healthy participants, men's and females aged from 18 up to 45 years inclusive;
3. Readiness of participants and their sexual partners to use reliable methods of contraception (a combination of at least two modes, including one barrier method, for example, use of a spermicide and condom) from the moment of signing of the informed consent (that is in 3 days before administration of drugs) and before the expiration of 1 month after completion of participation in the study;
4. The verified diagnosis "is healthy," established according to collecting the anamnesis and physical inspection:

   * absence in the anamnesis and at the time of screening clinically significant dysfunctions cardiovascular, respiratory, nervous, hemopoietic, endocrine, gastrointestinal systems, liver, and kidneys;
   * absence of persistent infections (HIV, hepatitis B, C, syphilis);
   * absence within 30 days before inclusion in the study of sharp, infectious diseases;
   * absence of the mental disorders and any other states capable to affectability of the participant to follow requirements of the protocol;
   * lack of complaints to the state of health within 30 days before inclusion in the study;
   * hemodynamic indicators within norm: systolic arterial blood pressure - within 100 - 130 mm Hg., diastolic arterial blood pressure - within 60 - 90 mm Hg;
5. The Body Mass Index (BMI) is in normal limits (≥18.5 kg/sq.m and ≤30 kg/sq.m);
6. There is a lack of instructions on alcohol abuse or narcotic dependence at the time of inclusion in study or the anamnesis;
7. The participant's Ability, according to the study, to fulfill the requirements of the protocol.

Exclusion Criteria:

1. The severe vaccine-challenged reactions/complications connected with the previous vaccination;
2. Allergic reactions to components of vaccine or any previous vaccination;
3. Any carried-out vaccination less than in 2 months before the present study;
4. In the chronic anamnesis diseases of the digestive tract, causes intestinal invagination, gastrointestinal pathology, surgical interventions on abdominal organs;
5. Clinically significant deviations of laboratory and tool indicators (including standard pathological changes on the ECG) overstepping the bounds of the range of normal values revealed on screening and capable of negatively impacting the safety of participants of the volunteer in the study;
6. Any diseases within four weeks preceding screening;
7. Presence of any oncological diseases (including in the anamnesis);
8. Any disease demands continuous therapy, including vegetable drugs or the expected concurrent therapy during the study;
9. Donor blood donation (450 ml of blood or plasma and more) or loss of 500 or more ml of blood in 3 months before the study;
10. Positive analysis on HIV, Hepatitis B and C, and syphilis (RW);
11. Impossibility to give the written informed consent or to follow requirements of the protocol;
12. Probability to refuse to follow the protocol's requirements, instructions and restrictions; for example, unwillingness to cooperate, impossibility to return to clinical center for the subsequent visits, and the probability not of completion of participation in a clinical trial;
13. Participation in clinical trials of drugs less than in 3 months before the study;
14. Smoking more than ten cigarettes in a day;
15. Drug addiction in the anamnesis. The positive analysis of urine on psychotropic and narcotic substances, psychoactive medicines;
16. Regular alcohol intake in many ˃10 units a week (to 1 unit of alcohol is equivalent to ½ l of beer, 200 ml of wine, or 50 ml of hard liquors) or anamnestic data on alcoholism. Alcohol intake within 48 hours before the Screening visit. Positive respiratory test for alcohol on screening (breathalyzer);
17. Observance of a special diet (for example, vegetarian, observance of a post, etc.) or lifestyle (including work at night and extreme physical activities, such as sport or raising of weights) which can interfere with carrying out the study;
18. The study cannot include military personnel or employees law enforcement agencies serving sentences in places of detention or being in custody;
19. The presence of conviction of the study is that the volunteer will not follow procedures of the protocol;
20. Use of any medicines, including OTC, vegetable medicines, dietary supplements, within 14 days before the study, according to the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Geometric Mean Titer (GMT) of antibody | 28 days post-Dose 1
Seroconversion level | 28 days after Dose 1 of vaccine
Seroconversion factor (The increase in the geometric mean antibody titer on day 28 compared to the initial level is expressed in the fold increase.). | 28 days post-Dose 1
  The seroconversion factor after administration of the study vaccine was 1.20, after administration of placebo - 0.97.
Frequency and expressiveness of AE /SAE. | From the time of Dose 1 to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Irina V. Feldblium, Dr. Sci, Study Director — Perm State Medical University named after Academician E.A. Wagner
Locations (1):
- Perm State Medical University named after Academician E.A. Wagner, Perm, Russia